CLINICAL TRIAL: NCT03650556
Title: Safety and Effectiveness of TactiCath™ Contact Force, Sensor Enabled™ (TactiCath SE) Catheter for Ablation of Drug Refractory, Symptomatic, Persistent Atrial Fibrillation (PERSIST-END IDE)
Brief Title: Safety and Effectiveness of TactiCath™ Contact Force, Sensor Enabled™ (TactiCath SE) Catheter for Ablation of Drug Refractory, Symptomatic, Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10239
Record Dates: First submitted 2018-08-01; First posted 2018-08-28 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ablation (Experimental): Enrolled subjects who had the investigational catheter inserted into their vasculature for pulmonary vein isolation by radiofrequency ablation treatment TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE).
  Interventions: Device: TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™

INTERVENTIONS:
Device: TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ — Ablation procedure for Persistent AF

SUMMARY:
This clinical investigation is intended to demonstrate the safety and effectiveness of the TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE) for use in cardiac electrophysiological mapping and for the treatment of drug-refractory, recurrent symptomatic persistent atrial fibrillation (AF) when used in conjunction with a compatible radiofrequency (RF) generator and three-dimensional mapping system. This clinical investigation will be conducted under an investigational device exemption (IDE) and is intended to support market approval of the TactiCath SE ablation catheter for the treatment of drug refractory, symptomatic persistent atrial fibrillation in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must provide written informed consent prior to any clinical investigation related procedure.
2. Documented symptomatic persistent AF, which is defined as continuous AF sustained beyond 7-days and less than 1-year that is documented by (1) a physician's note and (2) a 24-hour Holter within 90-days prior to the procedure, showing continuous AF
3. Refractory or intolerant to at least one Class I-IV antiarrhythmic drug (AAD) as evidenced by recurrent symptomatic AF
4. Age 18 years or older
5. Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

1. Continuous AF > 12 months (longstanding persistent AF)
2. Previous left atrial surgical or catheter ablation for atrial fibrillation or a previous procedure that required an incision in the left atrium with resulting scar
3. Any cardiac procedure (surgical or percutaneous) within 90-days prior to the initial procedure
4. CABG surgery within the 6-months (180-days) prior to the initial procedure
5. Valvular cardiac surgical/percutaneous procedure (i.e. ventriculotomy, valve repair or replacement and/or presence of a prosthetic or mechanical valve)
6. Any carotid stenting or endarterectomy
7. Documented or known left atrial thrombus on imaging
8. Left atrial diameter > 50 mm (parasternal long axis view or by CT)
9. Left ventricular ejection fraction < 40%
10. Unable to take anticoagulation medication due to contraindication or intolerance
11. History of blood clotting or bleeding abnormalities
12. Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI) within the 3-months (90-days) prior to the initial procedure
13. Documented thromboembolic event (including TIA) within the 12-months (365 days) prior to the initial procedure
14. Rheumatic heart disease
15. Uncontrolled heart failure or NYHA functional class III or IV
16. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2)
17. Awaiting cardiac transplantation or other cardiac surgery within the 12-months (365 days) following the initial ablation procedure
18. Unstable angina at the time of the initial procedure
19. Acute illness or active systemic infection or sepsis
20. AF secondary to electrolyte imbalance, thyroid disease, acute alcohol intoxication, major surgical procedure in the preceding 3-months, or other reversible or non-cardiac cause
21. Diagnosed atrial myxoma
22. Presence of implanted implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy-defibrillator (CRT-D)
23. Significant pulmonary disease, (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
24. Significant congenital anomaly or other anatomic or comorbid medical problem that in the opinion of the investigator would preclude enrollment in this study or compliance with the follow-up requirements or impact the scientific soundness of the clinical trial results
25. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period
26. Enrollment in an investigational study evaluating another device, biologic, or drug that may interfere with this clinical investigation at the time of the initial procedure or within 30 days prior to the initial procedure
27. Presence of any condition that precludes appropriate vascular access or manipulation of catheter
28. Life expectancy less than 12-months
29. Body mass index > 40 kg/m2
30. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
31. Renal failure requiring dialysis
32. Vulnerable subject
33. History of atriotomy or ventriotomy
34. Implanted endocardial left atrial appendage occlusion device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (20):
  - University Hospital (UAB), Birmingham, Alabama
  - St. Bernards, Jonesboro, Arkansas
  - Arkansas Heart Hosptial, Little Rock, Arkansas
  - Scripps Health, La Jolla, California
  - Sequoia Hospital, Redwood City, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - Florida Hospital, Orlando, Florida
  - Emory University Hosptial, Atlanta, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Jackson Heart Clinic, Jackson, Mississippi
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York University Hospital, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia, Austin, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital - City Campus, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A patient is considered enrolled from the moment the patient provides written informed consent and meets all eligibility criteria
Pre-assignment Details: One subject was withdrawn after meeting enrollment criteria but prior to procedure with the investigational device.
Groups:
- Enrolled: A patient is considered enrolled from the moment the patient provides written informed consent and meets all eligibility criteria
Period: Overall Study
Arm/Group | Enrolled
Started | 224
Ablation Procedure | 223
Pre-Discharge | 223
7-day Follow-Up | 223
3-month Follow-Up | 210
6-month Follow-up | 197
12-month Follow-Up | 189
15-month Follow-Up | 187
Completed | 187
Not Completed | 37
Not completed — Death | 2
Not completed — Withdrawal by Subject | 20
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 8
Not completed — Subject did not complete follow-up but did not meet criteria for lost-to-follow-up | 4
Not completed — Enrolled, but no ablation performed-investigational catheter was not inserted | 1

BASELINE CHARACTERISTICS:
Groups:
- Ablation: All enrolled subjects who had the investigational catheter inserted into their vasculature for pulmonary vein isolation by radiofrequency ablation treatment
Arm/Group | Ablation
Number analyzed (Participants) | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 209
  Unknown or Not Reported | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 213
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 209
  Australia | 14

OUTCOME MEASURES:

1. Primary Outcome: Rate of Subjects With a Device and/or Procedure-related SAE.
Description: Rate of subjects with a device and/or procedure-related SAE with onset within 7-days of any ablation procedure that used the investigational device.
Time Frame: Within 7 days of initial or repeat procedure performed ≤180 days of initial procedure
Population: The analysis population for the primary safety endpoint is all enrolled subjects who had the investigational catheter inserted into their vasculature for pulmonary vein isolation by radiofrequency ablation treatment and who have completed their 7-day follow-up visit; or crossed the end of the 7-day visit window without the visit but with a primary safety endpoint event
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 223
Participants | 7

2. Primary Outcome: Percent of Subjects Free From Atrial Fibrillation (AF), Atrial Flutter (AFL) or Atrial Tachycardia (AT) Recurrence.
Description: The following events were considered a failure for AF/AFL/AT recurrence:
  * If AF/AFL/AT recurrence (>30 second episode) occurred at any time after the therapy consolidation period (>180 days after the initial procedure), or
  * If the subject required a repeat procedure for the treatment of AF after the therapy consolidation period, the subject was considered an effectiveness endpoint failure regardless of documentation of a >30 second AF/AFL/AT episode, or
  * If the subject required a second repeat procedure at any time after the initial procedure, or
  * If the subject required a new AAD or a previously failed AAD at a dose greater than the highest ineffective historical dose for AF after the therapy consolidation period, or
  * If the subject required a cardioversion (electrical or pharmacological) for the treatment of AF after the therapy consolidation period, or
  * If the subject had a continuous atrial arrhythmia throughout a 12-lead ECG recording after the the
Time Frame: 15 months
Population: The analysis population for the primary effectiveness endpoint is all enrolled subjects who had the investigational catheter inserted into their vasculature for pulmonary vein isolation by radiofrequency ablation treatment and who have completed their 15-month ECG, TTM, and/or 24-hour Holter assessment; or crossed the end of the 15-month visit window without the ECG, TTM and/or 24-hour Holter assessment but with a prior primary effectiveness endpoint event.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 190
Participants | 114

3. Secondary Outcome: Acute Procedural Success
Description: Percent of subjects who achieve acute procedural success defined as confirmation of entrance block in all pulmonary veins
Time Frame: Immediate post procedure
Population: The analysis population is all enrolled subjects who had the investigational catheter inserted into their vasculature for pulmonary vein isolation by radiofrequency ablation treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 223
Participants | 219

4. Secondary Outcome: 15-month Success Off of Antiarrhythmic Drugs
Description: Percent of subjects off all AADs taken to treat AF/AFL/AT who achieve15-month success, defined as freedom from documented AF/AFL/AT recurrence (episodes >30 seconds) during the 9-month period following the blanking and therapy consolidation periods.
Time Frame: 15 months
Population: The analysis population is all enrolled subjects who had the investigational catheter inserted into their vasculature for pulmonary vein isolation by radiofrequency ablation treatment and who have completed their 15-month ECG, TTM, and/or 24-hour Holter assessment; or crossed the end of the 15-month visit window without the ECG, TTM and/or 24-hour Holter assessment but with a prior primary effectiveness endpoint event.
Measure: Count of Participants; unit: Participants
Groups:
- Ablation: Pulmonary vein isolation by radiofrequency ablation treatment TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™ (TactiCath SE) in the persistent AF population.
  TactiCath™ Contact Force Ablation Catheter, Sensor Enabled™: Ablation procedure for Persistent AF
Arm/Group | Ablation
Number analyzed (Participants) | 190
Participants | 89

5. Secondary Outcome: 15 Month Single Procedure Success
Description: Percent of subjects who achieve 15-month single procedure success, defined as freedom from documented AF/AFL/AT recurrence (episodes >30 seconds) during the 9-month period following the blanking and therapy consolidation periods after a single ablation procedure. Any repeat ablation procedure required by the subject at any time was deemed an effectiveness failure in this analysis.
Time Frame: 15 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ablation
Number analyzed (Participants) | 190
Participants | 110

ADVERSE EVENTS:
Time Frame: 15 months
Description: An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device under investigation.
Arm/Group | Enrolled
All-Cause Mortality (participants affected / at risk) | 2/224
Serious Adverse Events (participants affected / at risk) | 59/224
Other Adverse Events (participants affected / at risk) | 29/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled (N=224)
Arrhythmia (Cardiac disorders) | 9 (9)
Bleeding/Anemia (Vascular disorders) | 5 (5)
Cerebrovascular Accident/Stroke (Nervous system disorders) | 2 (3)
Coronary Artery Thrombosis/Occlusion (Cardiac disorders) | 1 (1)
Elective Procedure/Surgery (General disorders) | 5 (5)
Heart Failure/Pump Failure (Cardiac disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Infection (Infections and infestations) | 4 (4)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Decompensation/Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Respiratory Compromise/Decompensation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Shock (Vascular disorders) | 1 (1)
Syncope/Dizziness (General disorders) | 1 (1)
Valve Insufficiency (Cardiac disorders) | 1 (1)
Volume Overload (Vascular disorders) | 3 (3)
Acute Ischemic Colitis (Gastrointestinal disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Collapse (General disorders) | 1 (1)
Colon Obstruction (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fracture of Humerous (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower GI Bleed (Gastrointestinal disorders) | 2 (2)
Pelvic Inflammatory Disease (Infections and infestations) | 1 (1)
Penile Fracture (Reproductive system and breast disorders) | 1 (1)
Rectal and Vaginal Prolapse Repair (General disorders) | 1 (1)
Right Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Sick Sinus Symptom (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Sudden Cardiac Death (General disorders) | 1 (1)
Trauma (General disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Chest Pain/Discomfort (Cardiac disorders) | 8 (8)
Cardiac Perforation or Tamponade (Cardiac disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Encephalopathy (Psychiatric disorders) | 1 (1)
Jaw and Neck Pain (General disorders) | 1 (1)
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled (N=224)
Air Embolism (Injury, poisoning and procedural complications) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Chest Pain/Discomfort (Cardiac disorders) | 5 (5)
Infection (Infections and infestations) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/Thrombus (Blood and lymphatic system disorders) | 1 (1)
Transient Ischemic Attack (General disorders) | 1 (1)
Vascular Access Complication (Vascular disorders) | 2 (2)
Vascular Bleeding/Local Hematoma/Ecchymosis (Vascular disorders) | 5 (5)
Volume Overload (Vascular disorders) | 3 (3)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Cough (General disorders) | 2 (2)
Elevated Troponin (Blood and lymphatic system disorders) | 1 (1)
Esophageal Inflammation (Gastrointestinal disorders) | 1 (1)
Fluid Retention (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Hepatohepatomegaly With Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1)
Jaw Pain (General disorders) | 1 (1)
Shoulder Blade/ Arm Pit Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Trochanteric Bursitis (Blood and lymphatic system disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03650556/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03650556/SAP_002.pdf